CLINICAL TRIAL: NCT02408380
Title: Analysis of a Biomarker Signature, Consisting of Toll-like Receptor 2 (TLR2), TLR4 and CCR1, by Flow Cytometry in Patients With MS Treated With Gilenya (FTY720)
Brief Title: Analysis of a Biomarker Signature in Patients With Multiple Sclerosis (MS) Treated With Gilenya (FTY720)
Acronym: MS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Haegert, Doctor, McGill University
Other Study IDs: CFTY720DCA05T
Record Dates: First submitted 2015-03-20; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Sclerosis
Keywords: biomarker; disease progression
MeSH Terms: conditions — Multiple Sclerosis; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cryopreserved peripheral blood mononuclear cells.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study investigates whether there is a link between disease activity/progression in patients receiving Gilenya and expression of a putative biomarker signature in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Gilenya modulates expression of the sphingosine-1-phosphate receptor and inhibits egress of several lymphocyte subsets from lymph nodes. This results in immunosuppression that has a beneficial effect in patients with multiple sclerosis.

Our laboratory reported that increased expression of a possible biomarker signature, consisting of TLR2, TLR4 and CCR1, in a T-subset is associated with rapid MS progression. The investigators will test whether a significant proportion of patients at baseline upregulate this biomarker signature in one or more T-subsets, whether expression of this biomarker signature changes with treatment with Gilenya and whether expression levels of this signature predict disease activity or progression over a 12 month followup period. The investigators will study patients who are already being treated with Gilenya by their neurologists or who are already being treated with Gilenya as part of a clinical trial sponsored by Novartis Pharmaceuticals Canada. Patients will not be treated with Gilenya for the purposes of our study.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with Gilenya

Exclusion Criteria:

* Subject is under 18 or over 65.
* Subject has less than 4 weeks of discontinuation with steroid treatment for a relapse.
* Subject cannot communicate reliably with investigator.
* Vulnerable subjects exclude, namely patients defined as those without freedom by the law (e.g. prisoners or by administrative decision) or people hospitalized without their consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients treated with Gilenya compared with age-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in expression of a biomarker signature | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Haegert, MD, Principal Investigator — MUHC research institute
Locations (1):
- McGill University, Montreal, Quebec, Canada